CLINICAL TRIAL: NCT05487651
Title: Allogeneic Natural Killer T-Cells Expressing CD19 Specific Chimeric Antigen Receptor and Interleukin-15 in Relapsed or Refractory B-Cell Malignancies 2
Brief Title: Allogeneic NK T-Cells Expressing CD19 Specific CAR in B-Cell Malignancies
Acronym: ANCHOR2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATX-K502-001
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: NHL, Relapsed, Adult; B-cell Lymphoma; B-cell Leukemia; DLBCL - Diffuse Large B Cell Lymphoma; ALL, Adult B Cell; ALL, Childhood; CLL/SLL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Lymphoma, B-Cell; Leukemia, B-Cell; Dendritic Cell Sarcoma, Interdigitating; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A, non-ALL relapsed/refractory (Experimental): These dose levels will be evaluated. Patients will also receive lymphodepletion chemotherapy consisting of cyclophosphamide and fludarabine followed by CD19.CAR-aNKT cell infusion.
  Genetic: CD19.CAR-aNKT cells Patients will be given the T-cell product by intravenous injection (into the vein through an IV line) at the assigned dose.
  Dose level 1: 1×107/m2. Dose level 2: 3×107/m2. Dose level 3: 1×108/m2).
  Drug: Cyclophosphamide:
  Lymphodepletion chemotherapy. Patients will receive 3 daily doses of cyclophosphamide (500mg/m2/day finishing at least 24 hours before T-cell infusion. The drug will be given intravenously (through an IV needle) Other name: Cytoxan
  Drug Fludarabine Lymphodepletion chemotherapy. Patient will receive 3 daily dose of fludarabine (30mg/m2/day) finishing at least 24 hours before T-cell infusion. the drug will be given intravenously (through an IV needle) Other name: Fludara
  Interventions: Genetic: KUR-502
- Cohort B, ALL releapsed/refractory (Experimental): This cohort is for patients with relapsed or refractory B-cell ALL afer 2 or more lines of therapy. Patients will also receive lymphodepletion chemotherapy consisting of cyclophosphamide and fludarabine followed by the CD19.CAR-aNKT cell infusion.
  Genetic: CD19.CAR-aNKT cells Patients will be given the T-cell product by intravenous injection (into the vein through an IV line) at the assigned dose.
  Dose level 1: 1×107/m2. Dose level 2: 3×107/m2. Dose level 3: 1×108/m2).
  Drug: Cyclophosphamide:
  Lymphodepletion chemotherapy. Patients will receive 3 daily doses of cyclophosphamide (500mg/m2/day finishing at least 24 hours before T-cell infusion. The drug will be given intravenously (through an IV needle) Other name: Cytoxan
  Drug Fludarabine Lymphodepletion chemotherapy. Patient will receive 3 daily dose of fludarabine (30mg/m2/day) finishing at least 24 hours before T-cell infusion. the drug will be given intravenously (through an IV needle)
  Interventions: Genetic: KUR-502

INTERVENTIONS:
Genetic: KUR-502 — KUR-502 (CD19.CAR-aNKT cells) consists of transduced allogeneic natural killer T cells (aNKT) genetically modified with additional features to enhance their anti-tumor activity against CD19+ B-cell malignancies. Following intravenous (IV) infusion, the product is expected to kill CD19+ tumor cells by direct interaction with the chimeric antigen receptor (CAR), and activation of the NKT cells to kill tumor through their innate cell killing.
  Other Names: CD19.CAR-aNKT cells

SUMMARY:
This study is a multi-center study to evaluate the safety of KUR-502 in subjects with refractory/relapsed B-cell NHL or leukemia (ALL or CLL).

DETAILED DESCRIPTION:
KUR-502 will be manufactured from leukapheresis products from healthy donors. Subjects will be enrolled into 2 parallel cohorts (Cohort A [non-ALL] and Cohort B [ALL]). Each cohort will undergo dose escalation independently.

Three (3) dose levels will be evaluated in the ANCHOR and ANCHOR2 studies combined (1×107/m2, 3×107/m2, 1×108/m2). Dose levels are defined based on the number of transduced KUR-502 cells. Body surface area (BSA) will be capped at 2.4 m2. Subjects will receive <1×104 allogeneic T cells/kg at any dose level.

The MTD will be determined once dose escalation is completed, and all subjects are evaluable for DLT. If there is no DLT that determines an MTD, a maximum dose level will be declared. Dose escalation will stop when 6 subjects have been treated at the MTD or highest dose level.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects must meet all of the following criteria to be included in this study:

1. Signed written informed consent.
2. Diagnosis of CD19+ B-cell lymphoma or leukemia (ALL or CLL).

   * Subjects who previously received CD19-directed therapy must have biopsy or flow cytometry-confirmed CD19+ tumor following the CD19-directed therapy; may be performed by local laboratory.
3. The disease is:

   Cohort A (non-ALL subjects):
   * Relapsed or refractory after ≥2 lines of therapy, including a CD20 antibody, if an indolent lymphoma.
   * Relapsed or refractory after ≥2 lines of therapy, including ibrutinib and venetoclax, if CLL.
   * Relapsed or refractory after ≥2 lines of therapy, including a CD20 antibody and an anthracycline, and the subject is ineligible for autologous stem cell transplantation, if an aggressive or highly aggressive lymphoma.
   * Ineligibility for autologous stem cell transplantation includes non-responsive disease after salvage therapy and failure to mobilize stem cells for transplant.

   Cohort B (ALL subjects):
   * Relapsed or refractory after ≥2 lines of therapy.
4. Measurable disease by current criteria (Lugano criteria for lymphomas, IWG criteria for CLL, and detectable disease for ALL).
5. Age 3 to 75 years; subjects <18 years old will not be enrolled as the first subject on any dose level.
6. BSA ≤2.4 m2.
7. Bilirubin <2 times the upper limit of normal (ULN) (3 times if the subject has Gilbert syndrome).
8. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <5 times ULN.
9. Estimated glomerular filtration rate (GFR) ≥50 mL/min.
10. Pulse oximetry ≥90% on room air.
11. Karnofsky or Lansky score ≥70.
12. Recovered from the acute toxic effects of all prior chemotherapy based on the enrolling physician's assessment (if some effects of chemotherapy are expected to last long term, for example, residual neuropathy, anemia, or alopecia, subject is eligible if meets other eligibility criteria).
13. Life expectancy >12 weeks.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

1. Females who are breastfeeding or pregnant at Screening (as documented by a positive urine or serum pregnancy test; may be performed by local laboratory).
2. Females of childbearing potential who:

   * Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) through the Day 365 visit or for 30 days after study drug discontinuation.
   * Are currently abstinent, and do not agree to use a double-barrier method (as described above) or refrain from sexual activity through the Day 365 visit or for 30 days after study drug discontinuation.
   * Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive through the Day 365 visit or for 30 days after study drug discontinuation.
3. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception through the Day 365 visit or for 30 days after study drug discontinuation). No sperm donation is allowed through the Day 365 visit or for 30 days after study drug discontinuation.
4. Currently receiving any investigational agents or received any cellular therapies within the previous 6 weeks prior to the KUR-502 infusion.
5. History of Grade 2 to 4 GvHD.
6. History of hypersensitivity reactions to murine protein-containing products.
7. Active infection with human immunodeficiency virus (HIV) or human T cell lymphotropic virus (HTLV).
8. Active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
9. Uncontrolled active bacterial, fungal, or other viral infection.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) rate and grade of single dose of Kur-502 | 4 weeks post T cell infusion
  Incidence rate and the grade (severity) of dose-limiting toxicities (DLTs) based on adverse events (AEs) reported according to the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - OHSU - Knight Cancer Center, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided